CLINICAL TRIAL: NCT00482573
Title: Maternal-Fetal Monitoring of Patients With Rheumatic Heart Disease During Dental Procedure Under Local Anesthesia
Brief Title: Dental Anesthesia in Pregnant Women With Rheumatic Heart Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Noedir Stolf, Faculdade de Medicina da Universidade de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAPPesq 009/03
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Rheumatic Heart Disease; Pregnancy; Dental Caries
Keywords: Electrocardiography, ambulatory/methods; Blood Pressure monitoring, ambulatory/methods; Cardiotocography/methods; Dental restoration, permanent; Anesthesia, local /methods; Lidocaine; Vasoconstrictor Agents; Epinephrine; Pregnancy; Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease; Dental Caries | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group LE (Experimental): Seventeen (54.8%) patients, composed group LE, were randomly assigned for the infusion of 1.8 mL (one cartridge) by the modified anesthesia into the periodontal ligament (PDLm injection) of 2% lidocaine solution with epinephrine 1:100,000. Their ages were ranging from 18 to 44 years (mean:29.6), they were diagnosed as having rheumatic valve disease, in a functional class I or II according to classification of the NYHA. Gestation age ranged from 28 to 36 weeks (mean:31.8), and the BMI from 18.7 to 32.9 (mean:23.8) kg/m2. All the patients had the restauration done in their inferior premolar and/or molar teeth.
  Interventions: Procedure: Dental local anesthesia
- Group LNE (Active Comparator): Fourteen (45.2%) patients, composed group LNE, were randomly assigned for the infusion of 1.8 mL (one cartridge) by the modified anesthesia into the periodontal ligament (PDLm injection) of 2% lidocaine solution without epinephrine. Their ages were ranging from 22 to 33 years (mean:26.6), they were diagnosed as having rheumatic valve disease, in a functional class I or II according to classification of the NYHA. Gestation age ranged from 29 to 37 weeks (mean:32.1), and the BMI from 18.5 to 38.1 (mean:22.8) kg/m2. All the patients had the restauration done in their inferior premolar and/or molar teeth.
  Interventions: Procedure: Dental local anesthesia

INTERVENTIONS:
Procedure: Dental local anesthesia — * 2% lidocaine solution with epinephrine 1:100,000
  * infusion of 1,8 mL (one cartridge)
  * Technic: modified anesthesia of the periodontal ligament (PDLm injection) was performed applying The Wand II Computerized System (Milestone International)
  Other Names: Alphacaine® 2% with epinephrine 1:100,000 - DFL; - fab/man 06/2003 - val/exp 06/2005 - lot 0306D11 and; - fab/man 04/2004 - val/exp 04/2006 - lot 0404D05
  Arms: Group LE
Procedure: Dental local anesthesia — * 2% lidocaine solution without vasoconstrictor
  * infusion of 1,8 mL (one cartridge)
  * Technic: modified anesthesia of the periodontal ligament (PDLm injection) was performed applying The Wand II Computerized System (Milestone International)
  Other Names: Xylestesin® 2% without vasoconstrictor - Cristália; - fab/man 06/2003 - val/exp 06/2006 - lot 3062010
  Arms: Group LNE

SUMMARY:
The hemodynamic parameters of 31 pregnant women with rheumatic valve disease, undergoing restorative dentistry under local anesthesia with 2% solution of lidocaine, divided in two groups, with (Group LE) and without 1:100,000 epinephrine solution (Group LNE), were studied by 24-hour ambulatory electrocardiographic monitoring, intermittent blood pressure monitoring and continuous cardiotocography, during three standard time periods. A significant decrease in the values of maternal heart rate was seen during the procedure, in comparison with the other two time periods in the two groups, as well as, the occurrence of cardiac arrhythmia in 9 (29.1%) patients, being 7 (41.8%) of them in the group receiving epinephrine anesthesia. We conclude the use of 2% lidocaine in association with epinephrine proved safe during dental procedure in pregnant women with rheumatic valve disease.

DETAILED DESCRIPTION:
During pregnancy, the organic systems of a woman are subjected to physiological modifications consequential to hormonal, anatomic and metabolical alterations. The most significant modification in the circulatory system is an increased cardiac output from the first three months of gestation. Women with heart disease may present with severe complications during the gestational period, because of inappropriate adaptation of her body to this hemodynamic overload, even those patients who are thought to have an appropriate functional capacity during early pregnancy. There are scant studies in the literature on the effects of local anesthetics, with and without vasoconstrictor, used in dental procedures on the cardiovascular variables of pregnant women with valvar disease, as well as on their concepti. Driven by this shortage, we decided to have this subject studied, by assessing and analyzing cardiotocographic parameters, such as fetal heart rate (FHR), fetal motility(FM) and uterine contractions (UC), in addition to blood pressure (BP) and electrocardiographic variables, such as heart rate (HR) and extrasystoles (ES), in pregnant women with rheumatic valvar disease who undergo local anesthesia with lidocaine, with and without vasoconstrictor, during restorative dental procedure. For this, 31 rheumatic heart disease patients who were in their 28th to 37th week of gestation, had 24-hour ambulatory monitoring of their BP and Holter electrocardiography (Holter-ECG), and cardiotocography (CTG), performed during: (1) baseline - 60 minutes before the procedure for BP and Holter-ECG monitoring, and 20 minutes before the procedure for CTG; (2) procedure - 56±15.5 minutes (mean±SD); (3) post-procedure - 20 minutes; and (4) mean 24-hour HR and ES measurement, and mean wake and sleeping periods BP monitoring. Variation of the above variables was analyzed in two groups, one with infusion of a 2% solution of lidocaine without vasoconstrictor (Group LNE) composed of 14 patients, and the other with infusion of a 2% solution of lidocaine with epinephrine 1:100,000 (Group LE) composed of 17 patients, randomized drawing and single blind. The investigator wise person which solution of lidocaine was being used, therefore the proper local vasoconstriction denounced if it was infiltrated or not epinephrine. The used technique was of the modified periodontal ligament (PDLm injection), by means of the equipment The Wand, infusing 1.8 ml (one cartridge) in six minutes. We use the technique of analysis of variance (ANOVA) with repeated measures to calculate the size of the sample and for the analysis and multiple interpretation of the variable in three distinct periods, on the basis of the table of Vonesh and Shork (15 patients in each group, considering a correlation enters the measures of next value the 0,4, a level of significance of 5% and to be able of test of 80%). All the variable had been initially analyzed descriptive. For the quantitative variable this analysis was made through the comment of the minimum and maximum values, and of the calculation of medium averages and shunting line-standard and. For the qualitative variable we calculate absolute and relative frequencies. The level of significance used for the tests was of 5% (p<0,05).The maternal HR values obtained during the procedure showed a significant reduction only in comparison with the other time periods (P<0.001)in the two groups. The comparison of the groups LE e LNE did not reveal any significant difference (P>0.05). ES was detected in 9 (29.0%) patients, being 7 of them (41.8%) from the Group LE. BP did not show any significant difference neither between time periods, nor between groups (P>0.05). The same occurred in the comparative analysis of the fetal parameters obtained during CTG - number of UC, level and variability from baseline of the FHR, number of accelerations of the FHR and fetal reactivity pattern. Our conclusion was that the use of 2% solution of lidocaine in association with epinephrine proved safe during dental procedure in pregnant women with rheumatic valvar cardiopathy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria: women with rheumatic valvar disease as diagnosed by the clinical history and physical examination, and documented by Doppler echocardiography, either having undergone surgical or percutaneous intervention before becoming pregnant or not, in functional class (FC) I or II, according to classification of the New York Heart Association (NYHA).
* Obstetrical criteria: one fetus pregnancy, gestational age (GA) between 28 and 37 weeks.
* Odontological criteria: total or partial dentition, with the presence of lower premolar and/or molar teeth in need of restorative dentistry due to development of dental caries (Black Class I, II and/or V), or due to the presence of restorations with edge infiltration clinically and/or radiographically diagnosed recurrent caries.

Exclusion Criteria:

* Clinical criteria: heart failure, uncontrolled chronic arterial hypertension, or complex and/or symptomatic ventricular arrhythmia.
* Obstetrical criteria: preeclampsia, uterine growth restriction, and labor.
* Odontological criteria: dental caries in lower premolar or molar tooth with clinical and/or radiographic diagnosis of pulpal exposure, pulpitis, or pulpal necrosis, fracture or destruction of the tooth crown with prognostic of endodontic treatment or rehabilitation by prosthesis, or indication for extraction.
* Psychiatric criteria: patients with anxiety disorders such as panic, agoraphobia, social or specific phobias and obsessive-compulsive disorders, posttraumatic stress, or chemically-induced anxiety, according to the classification of the American Psychiatric Association (APA).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-04; Primary Completion 2005-07 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Maternal: Blood Pressure, Heart Rate and Extrasystoles; Maternal-Fetal: Fetal Heart Rate, number of uterine contractions, motility and fetal reactivity pattern, in function of presence or not of epinephrine 1:100000 in the 2% solution.of lidocaine | 4 periods Maternal: (1) Baseline - 60 minutes before the procedure, (2) Procedure, (3) Post-Procedure - 20 minutes, and (4) mean 24-hour; 3 periods Maternal-Fetal: (1) Baseline: 20 minutes before, (2) Procedure, and (3) Post-Procedure - idem maternal

SECONDARY OUTCOMES:
They had been the same analyses used for the Primary Outcome Measures, in function of the gestational age (GA): sub-group GA1 (15 pregnant women between 28 and 31 weeks) and sub-group GA2 (16 pregnant women between 28 and 31 weeks). | They had been the same periods established for the Time Frame of Primary Outcome Measure

CONTACTS AND LOCATIONS:
Overall Officials: Itamara LI Neves, PhD, Principal Investigator — Heart Institute (InCor) of University of São Paulo Medical School - Sao Paulo, Brazil
Locations (1):
- Heart Institute (InCor) of University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Dajani AS, Taubert KA, Wilson W, Bolger AF, Bayer A, Ferrieri P, Gewitz MH, Shulman ST, Nouri S, Newburger JW, Hutto C, Pallasch TJ, Gage TW, Levison ME, Peter G, Zuccaro G Jr. Prevention of bacterial endocarditis. Recommendations by the American Heart Association. Circulation. 1997 Jul 1;96(1):358-66. doi: 10.1161/01.cir.96.1.358. PMID 9236458
- [Background] Aellig WH, O'Neil R, Laurence DR, Verrill PJ. Cardiac effects of adrenaline and felypressin as vasoconstrictors in local anaesthesia for oral surgery under diazepam sedation. Br J Anaesth. 1970 Feb;42(2):174-6. doi: 10.1093/bja/42.2.174. No abstract available. PMID 5440531
- [Background] Ahn J, Pogrel MA. The effects of 2% lidocaine with 1:100,000 epinephrine on pulpal and gingival blood flow. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Feb;85(2):197-202. doi: 10.1016/s1079-2104(98)90426-7. PMID 9503456
- [Background] AKUTSU A, CHIBA T, TAKAHASHI H, SHIMODA M, SUEMATSU T. MANAGEMENT OF DENTAL PROBLEMS IN PATIENTS WITH CARDIOVASCULAR DISEASE. J Am Dent Assoc. 1964 Mar;68:333-42. doi: 10.14219/jada.archive.1964.0104. No abstract available. PMID 14128020
- [Background] Anwari JS, Butt AA, Al-Dar MA. Obstetric admissions to the intensive care unit. Saudi Med J. 2004 Oct;25(10):1394-9. PMID 15494809
- [Background] Asghar F, Kokab H. Evaluation and outcome of pregnancy complicated by heart disease. J Pak Med Assoc. 2005 Oct;55(10):416-9. PMID 16304847
- [Background] Assem ES, Punnia-Moorthy A. Allergy to local anaesthetics: an approach to definitive diagnosis. A review with an illustrative study. Br Dent J. 1988 Jan 23;164(2):44-7. doi: 10.1038/sj.bdj.4806337. No abstract available. PMID 2449232
- [Background] AXELROD J. Metabolism of epinephrine and other sympathomimetic amines. Physiol Rev. 1959 Oct;39:751-76. doi: 10.1152/physrev.1959.39.4.751. No abstract available. PMID 13795318
- [Background] Beller GA, Smith TW, Abelmann WH, Haber E, Hood WB Jr. Digitalis intoxication. A prospective clinical study with serum level correlations. N Engl J Med. 1971 May 6;284(18):989-97. doi: 10.1056/NEJM197105062841801. No abstract available. PMID 5553483
- [Background] Bennett JA, Riegel B, Bittner V, Nichols J. Validity and reliability of the NYHA classes for measuring research outcomes in patients with cardiac disease. Heart Lung. 2002 Jul-Aug;31(4):262-70. doi: 10.1067/mhl.2002.124554. PMID 12122390
- [Background] Brent RL. Commentary on JAMA article by Hujoel et al. Health Phys. 2005 Apr;88(4):379-81. doi: 10.1097/01.hp.0000152109.40007.35. PMID 15761300
- [Background] Bryant EE, Douglas BH, Ashburn AD. Circulatory changes following prolactin administration. Am J Obstet Gynecol. 1973 Jan 1;115(1):53-7. doi: 10.1016/0002-9378(73)90088-4. No abstract available. PMID 4344064
- [Background] Bush RK, Taylor SL, Holden K, Nordlee JA, Busse WW. Prevalence of sensitivity to sulfiting agents in asthmatic patients. Am J Med. 1986 Nov;81(5):816-20. doi: 10.1016/0002-9343(86)90351-7. PMID 3535492
- [Background] Capeless EL, Clapp JF. Cardiovascular changes in early phase of pregnancy. Am J Obstet Gynecol. 1989 Dec;161(6 Pt 1):1449-53. doi: 10.1016/0002-9378(89)90902-2. PMID 2603897
- [Background] Caruana P, Pateromichelakis S, Rood JP. The effects of adrenaline on lignocaine nerve block anaesthesia. J Dent. 1982 Jun;10(2):140-3. doi: 10.1016/s0300-5712(82)80008-0. No abstract available. PMID 6955323
- [Background] Cawson RA, Curson I, Whittington DR. The hazards of dental local anaesthetics. Br Dent J. 1983 Apr 23;154(8):253-8. doi: 10.1038/sj.bdj.4805046. No abstract available. PMID 6344891
- [Background] Cintron G, Medina R, Reyes AA, Lyman G. Cardiovascular effects and safety of dental anesthesia and dental interventions in patients with recent uncomplicated myocardial infarction. Arch Intern Med. 1986 Nov;146(11):2203-4. PMID 3778050
- [Background] Colman JM, Sermer M, Seaward PG, Siu SC. Congenital heart disease in pregnancy. Cardiol Rev. 2000 May-Jun;8(3):166-73. doi: 10.1097/00045415-200008030-00007. PMID 11174890
- [Background] Cox JL, Gardner MJ. Treatment of cardiac arrhythmias during pregnancy. Prog Cardiovasc Dis. 1993 Sep-Oct;36(2):137-78. doi: 10.1016/0033-0620(93)90005-x. No abstract available. PMID 8103603
- [Background] Cruz SS, Costa Mda C, Gomes Filho IS, Vianna MI, Santos CT. [Maternal periodontal disease as a factor associated with low birth weight]. Rev Saude Publica. 2005 Oct;39(5):782-7. doi: 10.1590/s0034-89102005000500013. Epub 2005 Oct 24. Portuguese. PMID 16254655
- [Background] Dajani A, Taubert K, Ferrieri P, Peter G, Shulman S. Treatment of acute streptococcal pharyngitis and prevention of rheumatic fever: a statement for health professionals. Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease of the Council on Cardiovascular Disease in the Young, the American Heart Association. Pediatrics. 1995 Oct;96(4 Pt 1):758-64. PMID 7567345
- [Background] Davenport ES, Williams CE, Sterne JA, Murad S, Sivapathasundram V, Curtis MA. Maternal periodontal disease and preterm low birthweight: case-control study. J Dent Res. 2002 May;81(5):313-8. doi: 10.1177/154405910208100505. PMID 12097443
- [Background] Davenport ES, Williams CE, Sterne JA, Sivapathasundram V, Fearne JM, Curtis MA. The East London Study of Maternal Chronic Periodontal Disease and Preterm Low Birth Weight Infants: study design and prevalence data. Ann Periodontol. 1998 Jul;3(1):213-21. doi: 10.1902/annals.1998.3.1.213. PMID 9722705
- [Background] De Kock M, Gautier P, Vandewalle F, Renotte MT. Digoxin enhances bupivacaine toxicity in rats. Reg Anesth. 1991 Sep-Oct;16(5):272-7. PMID 1958605
- [Background] Fagade OO, Oginni FO. Intra-operative pain perception in tooth extraction--possible causes. Int Dent J. 2005 Aug;55(4):242-6. doi: 10.1111/j.1875-595x.2005.tb00322.x. PMID 16167613
- [Background] Finder RL, Moore PA. Adverse drug reactions to local anesthesia. Dent Clin North Am. 2002 Oct;46(4):747-57, x. doi: 10.1016/s0011-8532(02)00018-6. PMID 12436829
- [Background] Fisher JD. New York Heart Association Classification. Arch Intern Med. 1972 May;129(5):836. No abstract available. PMID 5025908
- [Background] Frabetti L, Checchi L, Finelli K. Cardiovascular effects of local anesthesia with epinephrine in periodontal treatment. Quintessence Int. 1992 Jan;23(1):19-24. PMID 1631266
- [Background] Frazier DT, Narahashi T, Yamada M. The site of action and active form of local anesthetics. II. Experiments with quaternary compounds. J Pharmacol Exp Ther. 1970 Jan;171(1):45-51. No abstract available. PMID 5410937
- [Background] Gall H, Kaufmann R, Kalveram CM. Adverse reactions to local anesthetics: analysis of 197 cases. J Allergy Clin Immunol. 1996 Apr;97(4):933-7. doi: 10.1016/s0091-6749(96)80067-4. PMID 8655888
- [Background] Garrow JS, Webster J. Quetelet's index (W/H2) as a measure of fatness. Int J Obes. 1985;9(2):147-53. PMID 4030199
- [Background] Gei AF, Hankins GD. Cardiac disease and pregnancy. Obstet Gynecol Clin North Am. 2001 Sep;28(3):465-512. doi: 10.1016/s0889-8545(05)70214-x. PMID 11512497
- [Background] Gilson GJ, Samaan S, Crawford MH, Qualls CR, Curet LB. Changes in hemodynamics, ventricular remodeling, and ventricular contractility during normal pregnancy: a longitudinal study. Obstet Gynecol. 1997 Jun;89(6):957-62. doi: 10.1016/s0029-7844(97)85765-1. PMID 9170474
- [Background] Gortzak RA, Abraham-Inpijn L, Peters G. Non-invasive 27-hour blood pressure registration including dental checkups in some dental practices. Clin Prev Dent. 1992 Sep-Oct;14(5):5-10. PMID 1291186
- [Background] Gortzak RA, Stegeman A, Ten Brinke R, Peters G, Abraham-Inpijn L. Ambulant 24-hour blood pressure and heart rate of dentists. Am J Dent. 1995 Oct;8(5):242-4. PMID 8634159
- [Background] Haas DA. An update on local anesthetics in dentistry. J Can Dent Assoc. 2002 Oct;68(9):546-51. PMID 12366885
- [Background] Hainsworth R. Reflexes from the heart. Physiol Rev. 1991 Jul;71(3):617-58. doi: 10.1152/physrev.1991.71.3.617. No abstract available. PMID 2057525
- [Background] Hainsworth R, Ledsome JR, Carswell F. Reflex responses from aortic baroreceptors. Am J Physiol. 1970 Feb;218(2):423-9. doi: 10.1152/ajplegacy.1970.218.2.423. No abstract available. PMID 5412457
- [Background] Hartung WH. Epinephrine and related compounds: influence of structure on physiologic activity. Chem Rev 9:389-465, 1931.
- [Background] Hasse AL, Heng MK, Garrett NR. Blood pressure and electrocardiographic response to dental treatment with use of local anesthesia. J Am Dent Assoc. 1986 Oct;113(4):639-42. doi: 10.14219/jada.archive.1986.0245. PMID 2945853
- [Background] Heinonen OP, Slone D, Shapiro S. Birth defects and drugs in pregnancy. Massachussets: Littleton; 1977.
- [Background] Hibbard LT. Maternal mortality due to cardiac disease. Clin Obstet Gynecol. 1975 Sep;18(3):27-36. doi: 10.1097/00003081-197509000-00005. No abstract available. PMID 1157363
- [Background] HOLTER NJ. New method for heart studies. Science. 1961 Oct 20;134(3486):1214-20. doi: 10.1126/science.134.3486.1214. PMID 13908591
- [Background] Houston JB, Appleby RC, DeCounter L, Callaghan N, Funk DC. Effect of r-epinephrine-impregnated retraction cord on the cardiovascular system. J Prosthet Dent. 1970 Oct;24(4):373-6. doi: 10.1016/0022-3913(70)90077-6. No abstract available. PMID 4195839
- [Background] Hunter L, Hunter B. Oral and dental problems associated with pregnancy. Oral healthcare in pregnancy and infancy. London: Macmillan Press Ltd; 1997. p. 27-34.
- [Background] Jackson D, Chen AH, Bennett CR. Identifying true lidocaine allergy. J Am Dent Assoc. 1994 Oct;125(10):1362-6. doi: 10.14219/jada.archive.1994.0180. PMID 7844301
- [Background] Johnson R, Swartz MH. A simplified approach to electrocardiography. New York: Saunders Company; 1986. p. 72-8.
- [Background] Kaplan EL. Cardiovascular disease in dental practice. In: Kaplan EL, editor. Dallas: American Heart Association. 1986
- [Background] Katz R, Karliner JS, Resnik R. Effects of a natural volume overload state (pregnancy) on left ventricular performance in normal human subjects. Circulation. 1978 Sep;58(3 Pt 1):434-41. doi: 10.1161/01.cir.58.3.434. No abstract available. PMID 679433
- [Background] Kaufman E, LeResche L, Sommers E, Dworkin SF, Truelove EL. Intraligamentary anesthesia: a double-blind comparative study. J Am Dent Assoc. 1984 Feb;108(2):175-8. doi: 10.14219/jada.archive.1984.0434. PMID 6584488
- [Background] Kohase H, Umino M. Allergic reaction to epinephrine preparation in 2% lidocaine: two case reports. Anesth Prog. 2004;51(4):134-7. PMID 15675262
- [Background] Lands AM, Arnold A, McAuliff JP, Luduena FP, Brown TG Jr. Differentiation of receptor systems activated by sympathomimetic amines. Nature. 1967 May 6;214(5088):597-8. doi: 10.1038/214597a0. No abstract available. PMID 6036174
- [Background] Lands AM, Luduena FP, Buzzo HJ. Differentiation of receptors responsive to isoproterenol. Life Sci. 1967 Nov 1;6(21):2241-9. doi: 10.1016/0024-3205(67)90031-8. No abstract available. PMID 6060269
- [Background] Lieb R. Anxiety disorders: clinical presentation and epidemiology. Handb Exp Pharmacol. 2005;(169):405-32. doi: 10.1007/3-540-28082-0_14. PMID 16594266
- [Background] Lipp M, Dick W, Daublander M, Fuder H, Stanton-Hicks M. Exogenous and endogenous plasma levels of epinephrine during dental treatment under local anesthesia. Reg Anesth. 1993 Jan-Feb;18(1):6-12. PMID 8448101
- [Background] LITWIN MS, GLEW DH. MANAGEMENT OF DENTAL PROBLEMS IN PATIENTS WITH CARDIOVASCULAR DISEASE. JAMA. 1964 Mar 14;187:848-9. doi: 10.1001/jama.1964.03060240056014. No abstract available. PMID 14094326
- [Background] Lopez NJ, Da Silva I, Ipinza J, Gutierrez J. Periodontal therapy reduces the rate of preterm low birth weight in women with pregnancy-associated gingivitis. J Periodontol. 2005 Nov;76(11 Suppl):2144-53. doi: 10.1902/jop.2005.76.11-S.2144. PMID 16277587
- [Background] Lopez NJ, Smith PC, Gutierrez J. Higher risk of preterm birth and low birth weight in women with periodontal disease. J Dent Res. 2002 Jan;81(1):58-63. doi: 10.1177/002203450208100113. PMID 11820369
- [Background] Lopez NJ, Smith PC, Gutierrez J. Periodontal therapy may reduce the risk of preterm low birth weight in women with periodontal disease: a randomized controlled trial. J Periodontol. 2002 Aug;73(8):911-24. doi: 10.1902/jop.2002.73.8.911. PMID 12211502
- [Background] Lopez R. Periodontal disease, preterm birth and low birthweight. Evid Based Dent. 2005;6(4):90-1. doi: 10.1038/sj.ebd.6400361. No abstract available. PMID 16355236
- [Background] Louro PM, Fiori HH, Filho PL, Steibel J, Fiori RM. [Periodontal disease in pregnancy and low birth weight]. J Pediatr (Rio J). 2001 Jan-Feb;77(1):23-8. doi: 10.2223/jped.105. Portuguese. PMID 14647615
- [Background] Lue HC, Wu MH, Wang JK, Wu FF, Wu YN. Long-term outcome of patients with rheumatic fever receiving benzathine penicillin G prophylaxis every three weeks versus every four weeks. J Pediatr. 1994 Nov;125(5 Pt 1):812-6. doi: 10.1016/s0022-3476(94)70082-6. PMID 7965439
- [Background] Lue HC, Wu MH, Wang JK, Wu FF, Wu YN. Three- versus four-week administration of benzathine penicillin G: effects on incidence of streptococcal infections and recurrences of rheumatic fever. Pediatrics. 1996 Jun;97(6 Pt 2):984-8. PMID 8637787
- [Background] LUND A. Release of adrenaline and noradrenaline from the suprarenal gland. Acta Pharmacol Toxicol (Copenh). 1951;7(4):309-20. doi: 10.1111/j.1600-0773.1951.tb02872.x. No abstract available. PMID 14894245
- [Background] Mabie WC, DiSessa TG, Crocker LG, Sibai BM, Arheart KL. A longitudinal study of cardiac output in normal human pregnancy. Am J Obstet Gynecol. 1994 Mar;170(3):849-56. doi: 10.1016/s0002-9378(94)70297-7. PMID 8141215
- [Background] Malamed SF. Ação clínica de agentes específicos. In: Malamed SF, editor. Manual de anestesia local. Rio de Janeiro: Guanabara Koogan; 2001. p. 43-65.
- [Background] Malamed SF. Avaliação física e psicológica. In: Malamed SF, editor. Manual de anestesia local. Rio de Janeiro: Guanabara Koogan; 2001. p. 43-65.
- [Background] Malamed SF. Neurofisiologia. In: Malamed SF, editor. Manual de anestesia local. Rio de Janeiro: Guanabara Koogan; 2001. p. 43-65.
- [Background] Malamed SF. O tubete. In: Malamed SF, editor. Manual de anestesia local. Rio de Janeiro: Guanabara Koogan; 2001. p. 43-65.
- [Background] Malamed SF. Allergy and toxic reactions to local anesthetics. Dent Today. 2003 Apr;22(4):114-6, 118-21. No abstract available. PMID 12733413
- [Background] Mashini IS, Albazzaz SJ, Fadel HE, Abdulla AM, Hadi HA, Harp R, Devoe LD. Serial noninvasive evaluation of cardiovascular hemodynamics during pregnancy. Am J Obstet Gynecol. 1987 May;156(5):1208-13. doi: 10.1016/0002-9378(87)90146-3. PMID 3578440
- [Background] Mather LE, Long GJ, Thomas J. The binding of bupivacaine to maternal and foetal plasma proteins. J Pharm Pharmacol. 1971 May;23(5):359-65. doi: 10.1111/j.2042-7158.1971.tb09927.x. No abstract available. PMID 4396980
- [Background] Mazhar SB, Gul-e-Irum. Fetomaternal outcome in pregnancy with cardiac disease. J Coll Physicians Surg Pak. 2005 Aug;15(8):476-80. PMID 16202358
- [Background] Meadows M. Pregnancy and the drug dilemma. FDA Consum. 2001 May-Jun;35(3):16-20. No abstract available. PMID 11458544
- [Background] Meiller TF, Overholser CD, Kutcher MJ, Bennett R. Blood pressure fluctuations in hypertensive patients during oral surgery. J Oral Maxillofac Surg. 1983 Nov;41(11):715-8. doi: 10.1016/0278-2391(83)90187-8. PMID 6579257
- [Background] Menezes Ada S Jr, Moreira HG, Daher MT. Analysis of heart rate variability in hypertensive patients before and after treatment with angiotensin II-converting enzyme inhibitors. Arq Bras Cardiol. 2004 Aug;83(2):169-72; 165-8. Epub 2004 Aug 17. English, Portuguese. PMID 15322659
- [Background] Meral G, Tasar F, Sayin F, Saysel M, Kir S, Karabulut E. Effects of lidocaine with and without epinephrine on plasma epinephrine and lidocaine concentrations and hemodynamic values during third molar surgery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Aug;100(2):e25-30. doi: 10.1016/j.tripleo.2005.03.031. PMID 16037765
- [Background] Montoya ME, Karnath BM, Ahmad M. Endocarditis during pregnancy. South Med J. 2003 Nov;96(11):1156-7. doi: 10.1097/01.SMJ.0000054503.18393.1E. PMID 14632369
- [Background] Moreu G, Tellez L, Gonzalez-Jaranay M. Relationship between maternal periodontal disease and low-birth-weight pre-term infants. J Clin Periodontol. 2005 Jun;32(6):622-7. doi: 10.1111/j.1600-051X.2005.00722.x. PMID 15882221
- [Background] Morrow LA, Linares OA, Hill TJ, Sanfield JA, Supiano MA, Rosen SG, Halter JB. Age differences in the plasma clearance mechanisms for epinephrine and norepinephrine in humans. J Clin Endocrinol Metab. 1987 Sep;65(3):508-11. doi: 10.1210/jcem-65-3-508. PMID 3624412
- [Background] Narahashi T, Frazier T, Yamada M. The site of action and active form of local anesthetics. I. Theory and pH experiments with tertiary compounds. J Pharmacol Exp Ther. 1970 Jan;171(1):32-44. No abstract available. PMID 5410936
- [Background] Neville BW, Damm DD, Alen CMA,Bouquot JE. Patologia oral & Maxilo facial. Rio de Janeiro: Guanabara Koogan; 1998.
- [Background] Newman MG, Takei HH, Carranza FA. Periodontia clínica. 9ª ed. Rio de Janeiro: Guanabara Koogan; 2004.
- [Background] Niwa H, Sato Y, Matsuura H. Safety of dental treatment in patients with previously diagnosed acute myocardial infarction or unstable angina pectoris. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Jan;89(1):35-41. doi: 10.1016/s1079-2104(00)80011-6. PMID 10630939
- [Background] Niwa H, Satoh Y, Matsuura H. Cardiovascular responses to epinephrine-containing local anesthetics for dental use: a comparison of hemodynamic responses to infiltration anesthesia and ergometer-stress testing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Aug;90(2):171-81. doi: 10.1067/moe.2000.107534. PMID 10936836
- [Background] Niwa H, Sugimura M, Satoh Y, Tanimoto A. Cardiovascular response to epinephrine-containing local anesthesia in patients with cardiovascular disease. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Dec;92(6):610-6. doi: 10.1067/moe.2001.118903. PMID 11740477
- [Background] USE OF epinephrine in connection with procaine in dental procedures. J Am Med Assoc. 1955 Mar 5;157(10):854. No abstract available. PMID 13233041
- [Background] Nusstein J, Burns Y, Reader A, Beck M, Weaver J. Injection pain and postinjection pain of the palatal-anterior superior alveolar injection, administered with the Wand Plus system, comparing 2% lidocaine with 1:100,000 epinephrine to 3% mepivacaine. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Feb;97(2):164-72. doi: 10.1016/j.tripleo.2003.09.012. PMID 14970775
- [Background] Nusstein J, Reader A, Beck FM. Anesthetic efficacy of different volumes of lidocaine with epinephrine for inferior alveolar nerve blocks. Gen Dent. 2002 Jul-Aug;50(4):372-5; quiz 376-7. PMID 12640855
- [Background] Offenbacher S, Lieff S, Boggess KA, Murtha AP, Madianos PN, Champagne CM, McKaig RG, Jared HL, Mauriello SM, Auten RL Jr, Herbert WN, Beck JD. Maternal periodontitis and prematurity. Part I: Obstetric outcome of prematurity and growth restriction. Ann Periodontol. 2001 Dec;6(1):164-74. doi: 10.1902/annals.2001.6.1.164. PMID 11887460
- [Background] Oliver G, Schafer EA. The Physiological Effects of Extracts of the Suprarenal Capsules. J Physiol. 1895 Jul 18;18(3):230-76. doi: 10.1113/jphysiol.1895.sp000564. No abstract available. PMID 16992252
- [Background] Pallasch TJ. Vasoconstrictors and the heart. J Calif Dent Assoc. 1998 Sep;26(9):668-73, 676. PMID 9879236
- [Background] Patterson R, Anderson J. Allergic reactions to drugs and biologic agents. JAMA. 1982 Nov 26;248(20):2637-45. No abstract available. PMID 7143626
- [Background] Poppas A, Shroff SG, Korcarz CE, Hibbard JU, Berger DS, Lindheimer MD, Lang RM. Serial assessment of the cardiovascular system in normal pregnancy. Role of arterial compliance and pulsatile arterial load. Circulation. 1997 May 20;95(10):2407-15. doi: 10.1161/01.cir.95.10.2407. PMID 9170404
- [Background] Poppers PJ. Evaluation of local anaesthetic agents for regional anaesthesia in obstetrics. Br J Anaesth. 1975 Feb;47 suppl:322-7. PMID 1148108
- [Background] PRITCHARD JA. CHANGES IN THE BLOOD VOLUME DURING PREGNANCY AND DELIVERY. Anesthesiology. 1965 Jul-Aug;26:393-9. doi: 10.1097/00000542-196507000-00004. No abstract available. PMID 14313451
- [Background] Ray P, Murphy GJ, Shutt LE. Recognition and management of maternal cardiac disease in pregnancy. Br J Anaesth. 2004 Sep;93(3):428-39. doi: 10.1093/bja/aeh194. Epub 2004 Jun 11. PMID 15194627
- [Background] Ritchie JM, Greene NM. Anestésicos locais. In: Gilman AG,Goodman LS, Rall TW, Murad F, editors. As bases farmacológicas da terapêutica. 7ª ed. Rio de Janeiro: Editora Guanabara; 1987. p. 198-210.
- [Background] Ritchie JM, Ritchie B, Greengard P. The active structure of local anesthetics. J Pharmacol Exp Ther. 1965 Oct;150(1):152-9. No abstract available. PMID 5853695
- [Background] Ritchie JM, Ritchie B, Greengard P. The effect of the nerve sheath on the action of local anesthetics. J Pharmacol Exp Ther. 1965 Oct;150(1):160-4. No abstract available. PMID 5853696
- [Background] Roberts DH, Sowray JH. Local analgesia in dentistry. 3rd ed. Bristol: Harcourt Publishers Ltd; 1987. 192 p.
- [Background] Roberts GJ, Simmons NB, Longhurst P, Hewitt PB. Bacteraemia following local anaesthetic injections in children. Br Dent J. 1998 Sep 26;185(6):295-8. doi: 10.1038/sj.bdj.4809795. PMID 9803037
- [Background] Rogers MC. Principles and practice of anesthesiology. St. Louis: Mosby; 1993.
- [Background] Rogers SN. Dental attendance in a sample of pregnant women in Birmingham, UK. Community Dent Health. 1991 Dec;8(4):361-8. PMID 1790481
- [Background] Rood JP. Adverse reaction to dental local anaesthetic injection--'allergy' is not the cause. Br Dent J. 2000 Oct 14;189(7):380-4. doi: 10.1038/sj.bdj.4800776. PMID 11081949
- [Background] Rood JP. Local analgesia during pregnancy. Dent Update. 1981 Oct;8(7):483-5. No abstract available. PMID 6951785
- [Background] Rood JP, Cannell H. Plasma levels of lignocaine after peri-oral injections of two different concentrations. Pharmacol Ther Dent. 1978;3(1):45-7. PMID 273933
- [Background] Rood JP, Pateromichelakis S, Prokopiou AA. The effects of adrenaline on lignocaine anaesthesia of the isolated nerve. J Dent. 1982 Dec;10(4):342-5. doi: 10.1016/0300-5712(82)90029-x. No abstract available. PMID 6962213
- [Background] Rosivack RG, Koenigsberg SR, Maxwell KC. An analysis of the effectiveness of two topical anesthetics. Anesth Prog. 1990 Nov-Dec;37(6):290-2. PMID 2097909
- [Background] Rubler S, Damani PM, Pinto ER. Cardiac size and performance during pregnancy estimated with echocardiography. Am J Cardiol. 1977 Oct;40(4):534-40. doi: 10.1016/0002-9149(77)90068-6. No abstract available. PMID 910718
- [Background] Sachs BP, Brown DA, Driscoll SG, Schulman E, Acker D, Ransil BJ, Jewett JF. Hemorrhage, infection, toxemia, and cardiac disease, 1954-85: causes for their declining role in maternal mortality. Am J Public Health. 1988 Jun;78(6):671-5. doi: 10.2105/ajph.78.6.671. PMID 3369599
- [Background] Sadaniantz A, Kocheril AG, Emaus SP, Garber CE, Parisi AF. Cardiovascular changes in pregnancy evaluated by two-dimensional and Doppler echocardiography. J Am Soc Echocardiogr. 1992 May-Jun;5(3):253-8. doi: 10.1016/s0894-7317(14)80345-3. PMID 1622616
- [Background] Sadler L, McCowan L, White H, Stewart A, Bracken M, North R. Pregnancy outcomes and cardiac complications in women with mechanical, bioprosthetic and homograft valves. BJOG. 2000 Feb;107(2):245-53. doi: 10.1111/j.1471-0528.2000.tb11696.x. PMID 10688509
- [Background] Schmaltz AA, Neudorf U, Winkler UH. Outcome of pregnancy in women with congenital heart disease. Cardiol Young. 1999 Jan;9(1):88-96. doi: 10.1017/s1047951100007496. PMID 10323550
- [Background] Seng GF, Gay BJ. Dangers of sulfites in dental local anesthetic solutions: warning and recommendations. J Am Dent Assoc. 1986 Nov;113(5):769-70. doi: 10.14219/jada.archive.1986.0263. No abstract available. PMID 3465791
- [Background] Seng GF, Kraus K, Cartwright G, Nerone R, Pacione R. Confirmed allergic reactions to amide local anesthetics. Gen Dent. 1996 Jan-Feb;44(1):52-4. PMID 8940570
- [Background] Setnikar I. Ionization of bases with limited solubility. Investigation of substances with local anesthetic activity. J Pharm Sci. 1966 Nov;55(11):1190-5. doi: 10.1002/jps.2600551104. No abstract available. PMID 5969769
- [Background] Sindel LJ, deShazo RD. Accidents resulting from local anesthetics. True or false allergy? Clin Rev Allergy. 1991 Fall-Winter;9(3-4):379-95. doi: 10.1007/BF02802315. No abstract available. PMID 1782629
- [Background] Smith C. Pharmacology of local anaesthetic agents. Br J Hosp Med. 1994 Nov 2-15;52(9):455-60. PMID 7874360
- [Background] Strichartz G. Molecular mechanisms of nerve block by local anesthetics. Anesthesiology. 1976 Oct;45(4):421-41. doi: 10.1097/00000542-197610000-00012. PMID 9844
- [Background] Sveen K. Effect of the addition of a vasoconstrictor to local anesthetic solution on operative and postoperative bleeding, analgesia and wound healing. Int J Oral Surg. 1979 Aug;8(4):301-6. doi: 10.1016/s0300-9785(79)80052-6. PMID 120334
- [Background] Tagger E, Tagger M, Sarnat H, Mass E. Periodontal ligament injection in the dog primary dentition: spread of local anaesthetic solution. Int J Paediatr Dent. 1994 Sep;4(3):159-66. doi: 10.1111/j.1365-263x.1994.tb00125.x. PMID 7811670
- [Background] Tagger M, Tagger E, Sarnat H. Periodontal ligament injection: spread of the solution in the dog. J Endod. 1994 Jun;20(6):283-7. doi: 10.1016/s0099-2399(06)80817-4. PMID 7931025
- [Background] Tarasoutchi F, Spina GS. Profilaxia da febre reumática. Rev Soc Cardiol Estado de São Paulo 15(1): 85-91, 2005.
- [Background] Teerlink JR, Foster E. Valvular heart disease in pregnancy. A contemporary perspective. Cardiol Clin. 1998 Aug;16(3):573-98, x. doi: 10.1016/s0733-8651(05)70032-1. PMID 9742331
- [Background] Thomson PD, Melmon KL, Richardson JA, Cohn K, Steinbrunn W, Cudihee R, Rowland M. Lidocaine pharmacokinetics in advanced heart failure, liver disease, and renal failure in humans. Ann Intern Med. 1973 Apr;78(4):499-508. doi: 10.7326/0003-4819-78-4-499. No abstract available. PMID 4694036
- [Background] Tucker GT. Plasma binding and disposition of local anesthetics. Int Anesthesiol Clin. 1975 Winter;13(4):33-59. doi: 10.1097/00004311-197513040-00005. No abstract available. PMID 1348
- [Background] Vanderheyden PJ, Williams RA, Sims TN. Assessment of ST segment depression in patients with cardiac disease after local anesthesia. J Am Dent Assoc. 1989 Sep;119(3):407-12. doi: 10.14219/jada.archive.1989.0048. PMID 2527898
- [Background] VERNALE CA. Cardiovascular responses to local dental anesthesia with epinephrine in normotensive and hypertensive subjects. Oral Surg Oral Med Oral Pathol. 1960 Aug;13:942-52. doi: 10.1016/0030-4220(60)90037-2. No abstract available. PMID 13841864
- [Background] Walton RE, Garnick JJ. The periodontal ligament injection: histologic effects on the periodontium in monkeys. J Endod. 1982 Jan;8(1):22-6. doi: 10.1016/S0099-2399(82)80312-9. No abstract available. PMID 6948904
- [Background] Weiner N, Taylor P. Transmissão neuro-humoral: sistemas nervosos autônomo e motor somático. In: Gilman AG, Goodman LS,Rall TW, Murad F, editors. As bases farmacológicas da terapêutica. 7ª ed. Rio de Janeiro: Guanabara Koogan; 1987. p. 43-65.
- [Background] West GA, Reid KH, Bastawi AE. Autonomic responses to dental procedures in pedodontic patients during a standard restoration session. J Dent Res. 1983 Jun;62(6):728-32. doi: 10.1177/00220345830620060801. PMID 6343440
- [Background] Wildsmith JA, Tucker GT, Cooper S, Scott DB, Covino BG. Plasma concentrations of local anaesthetics after interscalene brachial plexus block. Br J Anaesth. 1977 May;49(5):461-6. doi: 10.1093/bja/49.5.461. PMID 861114
- [Background] Yagiela JA. Local anesthetics: a century of progress. Anesth Prog. 1985 Mar-Apr;32(2):47-56. PMID 2408504
- [Background] Yagiela JA. Vasoconstrictor agents for local anesthesia. Anesth Prog. 1995;42(3-4):116-20. No abstract available. PMID 8934977
- [Result] ACOG practice bulletin. Antepartum fetal surveillance. Number 9, October 1999 (replaces Technical Bulletin Number 188, January 1994). Clinical management guidelines for obstetrician-gynecologists. Int J Gynaecol Obstet. 2000 Feb;68(2):175-85. PMID 10717828
- [Result] Electronic fetal heart rate monitoring: research guidelines for interpretation. National Institute of Child Health and Human Development Research Planning Workshop. Am J Obstet Gynecol. 1997 Dec;177(6):1385-90. PMID 9423739
- [Result] Status report: the periodontal ligament injection. Council on Dental Materials, Instruments, and Equipment. J Am Dent Assoc. 1983 Feb;106(2):222-4. No abstract available. PMID 6572678
- [Result] Avila WS, Rossi EG, Ramires JA, Grinberg M, Bortolotto MR, Zugaib M, da Luz PL. Pregnancy in patients with heart disease: experience with 1,000 cases. Clin Cardiol. 2003 Mar;26(3):135-42. doi: 10.1002/clc.4960260308. PMID 12685620
- [Result] Aberg G. Studies on the duration of local anesthesia: a possible mechanism for the prolonging effect of "vasoconstrictors" on the duration of infiltration anesthesia. Int J Oral Surg. 1980 Apr;9(2):144-7. doi: 10.1016/s0300-9785(80)80051-2. PMID 6773898
- [Result] Abraham-Inpijn L, Borgmeijer-Hoelen A, Gortzak RA. Changes in blood pressure, heart rate, and electrocardiogram during dental treatment with use of local anesthesia. J Am Dent Assoc. 1988 Apr;116(4):531-6. doi: 10.14219/jada.archive.1988.0318. PMID 3164019
- [Result] BADER RA, BADER ME, ROSE DF, BRAUNWALD E. Hemodynamics at rest and during exercise in normal pregnancy as studies by cardiac catheterization. J Clin Invest. 1955 Oct;34(10):1524-36. doi: 10.1172/JCI103205. No abstract available. PMID 13263433
- [Result] Beck FM, Weaver JM 2nd. Blood pressure and heart rate responses to anticipated high-stress dental treatment. J Dent Res. 1981 Jan;60(1):26-9. doi: 10.1177/00220345810600010501. PMID 6934188
- [Result] Bhatla N, Lal S, Behera G, Kriplani A, Mittal S, Agarwal N, Talwar KK. Cardiac disease in pregnancy. Int J Gynaecol Obstet. 2003 Aug;82(2):153-9. doi: 10.1016/s0020-7292(03)00159-0. PMID 12873775
- [Result] Biehl D, Shnider SM, Levinson G, Callender K. Placental transfer of lidocaine: effects of fetal acidosis. Anesthesiology. 1978 Jun;48(6):409-12. doi: 10.1097/00000542-197806000-00006. PMID 27131
- [Result] Blinder D, Shemesh J, Taicher S. Electrocardiographic changes in cardiac patients undergoing dental extractions under local anesthesia. J Oral Maxillofac Surg. 1996 Feb;54(2):162-5; discussion 165-6. doi: 10.1016/s0278-2391(96)90438-3. PMID 8604063
- [Result] Blinder D, Manor Y, Shemesh J, Taicher S. Electrocardiographic changes in cardiac patients having dental extractions under a local anesthetic containing a vasopressor. J Oral Maxillofac Surg. 1998 Dec;56(12):1399-402; discussion 1402-3. doi: 10.1016/s0278-2391(98)90403-7. PMID 9846537
- [Result] Brand HS, Gortzak RA, Abraham-Inpijn L. Anxiety and heart rate correlation prior to dental checkup. Int Dent J. 1995 Dec;45(6):347-51. PMID 8666460
- [Result] Brand HS, Gortzak RA, Palmer-Bouva CC, Abraham RE, Abraham-Inpijn L. Cardiovascular and neuroendocrine responses during acute stress induced by different types of dental treatment. Int Dent J. 1995 Feb;45(1):45-8. PMID 7607744
- [Result] Braunwald E, Bloodwell RD, Goldberg LI, Morrow AG. STUDIES ON DIGITALIS. IV. OBSERVATIONS IN MAN ON THE EFFECTS OF DIGITALIS PREPARATIONS ON THE CONTRACTILITY OF THE NON-FAILING HEART AND ON TOTAL VASCULAR RESISTANCE. J Clin Invest. 1961 Jan;40(1):52-9. doi: 10.1172/JCI104236. No abstract available. PMID 16695846
- [Result] Brooks VL, Kane CM, Van Winkle DM. Altered heart rate baroreflex during pregnancy: role of sympathetic and parasympathetic nervous systems. Am J Physiol. 1997 Sep;273(3 Pt 2):R960-6. doi: 10.1152/ajpregu.1997.273.3.R960. PMID 9321874
- [Result] Buckley JA, Ciancio SG, McMullen JA. Efficacy of epinephrine concentration in local anesthesia during periodontal surgery. J Periodontol. 1984 Nov;55(11):653-7. doi: 10.1902/jop.1984.55.11.653. PMID 6594502
- [Result] Cannell H, Kerawala C, Webster K, Whelpton R. Are intraligamentary injections intravascular? Br Dent J. 1993 Oct 23;175(8):281-4. doi: 10.1038/sj.bdj.4808302. PMID 8217423
- [Result] Cannell H, Walters H, Beckett AH, Saunders A. Circulating levels of lignocaine after peri-oral injections. Br Dent J. 1975 Feb 4;138(3):87-93. doi: 10.1038/sj.bdj.4803383. No abstract available. PMID 1053919
- [Result] Cioffi GA, Chernow B, Glahn RP, Terezhalmy GT, Lake CR. The hemodynamic and plasma catecholamine responses to routine restorative dental care. J Am Dent Assoc. 1985 Jul;111(1):67-70. doi: 10.14219/jada.archive.1985.0038. PMID 3861687
- [Result] Clark S, Hofmeyr GJ, Coats AJ, Redman CW. Ambulatory blood pressure monitoring during pregnancy: validation of the TM-2420 monitor. Obstet Gynecol. 1991 Jan;77(1):152-5. PMID 1984216
- [Result] Corah NL. Development of a dental anxiety scale. J Dent Res. 1969 Jul-Aug;48(4):596. doi: 10.1177/00220345690480041801. No abstract available. PMID 5256508
- [Result] Danzell JD. Pregnancy and pre-existing heart disease. J La State Med Soc. 1998 Feb;150(2):97-102. PMID 9510617
- [Result] Davenport RE, Porcelli RJ, Iacono VJ, Bonura CF, Mallis GI, Baer PN. Effects of anesthetics containing epinephrine on catecholamine levels during periodontal surgery. J Periodontol. 1990 Sep;61(9):553-8. doi: 10.1902/jop.1990.61.9.553. PMID 2213464
- [Result] Dawes GS, Moulden M, Redman CW. Criteria for the design of fetal heart rate analysis systems. Int J Biomed Comput. 1990 May;25(4):287-94. doi: 10.1016/0020-7101(90)90032-p. PMID 2365491
- [Result] Defosse O. [Local anesthesia with and without vasoconstrictors: indications, contra-indications and complications in relation to the health of the patient]. Rev Belge Med Dent (1984). 1999;54(4):242-58. French. PMID 12723166
- [Result] Druzin ML, Fox A, Kogut E, Carlson C. The relationship of the nonstress test to gestational age. Am J Obstet Gynecol. 1985 Oct 15;153(4):386-9. doi: 10.1016/0002-9378(85)90075-4. PMID 3901768
- [Result] Edmondson HD, Roscoe B, Vickers MD. Biochemical evidence of anxiety in dental patients. Br Med J. 1972 Oct 7;4(5831):7-9. doi: 10.1136/bmj.4.5831.7. PMID 5078436
- [Result] Elkayam U, Bitar F. Valvular heart disease and pregnancy part I: native valves. J Am Coll Cardiol. 2005 Jul 19;46(2):223-30. doi: 10.1016/j.jacc.2005.02.085. PMID 16022946
- [Result] Evertson LR, Gauthier RJ, Schifrin BS, Paul RH. Antepartum fetal heart rate testing. I. Evolution of the nonstress test. Am J Obstet Gynecol. 1979 Jan 1;133(1):29-33. doi: 10.1016/0002-9378(79)90406-x. PMID 760532
- [Result] Friedman MJ, Hochman MN. A 21st century computerized injection system for local pain control. Compend Contin Educ Dent. 1997 Oct;18(10):995-1000, 1002-3; quiz 1004. PMID 9533309
- [Result] Galili D, Kaufman E, Garfunkel AA, Michaeli Y. Intraligamentary anesthesia--a histological study. Int J Oral Surg. 1984 Dec;13(6):511-6. doi: 10.1016/s0300-9785(84)80022-8. PMID 6439659
- [Result] Garcia G, Kuhn J. Curso intensivo teórico-prático de cardiotocografia. Course's manual, 150p. 2004.
- [Result] Gauthier RJ, Evertson LR, Paul RH. Antepartum fetal heart rate testing. II. Intrapartum fetal heart rate observation and newborn outcome following a positive contraction stress test. Am J Obstet Gynecol. 1979 Jan 1;133(1):34-9. PMID 760533
- [Result] Giuliani M, Grossi GB, Pileri M, Lajolo C, Casparrini G. Could local anesthesia while breast-feeding be harmful to infants? J Pediatr Gastroenterol Nutr. 2001 Feb;32(2):142-4. doi: 10.1097/00005176-200102000-00009. PMID 11321382
- [Result] Goldstein MA, Michelson EL, Dreifus LS. The electrocardiogram in valvular heart disease. Cardiovasc Clin. 1993;23:55-64. No abstract available. PMID 8416131
- [Result] Gortzak RA, Abraham-Inpijn L. Blood pressure measurements during dental checkups representative of 26-hour registration. Oral Surg Oral Med Oral Pathol. 1990 Dec;70(6):730-3. doi: 10.1016/0030-4220(90)90009-h. PMID 2263330
- [Result] Gortzak RA, Abraham-Inpijn L. Pain-induced hypertensive episode in the dental office. Gen Dent. 1995 May-Jun;43(3):274-6. No abstract available. PMID 8940586
- [Result] Gortzak RA, Abraham-Inpijn L, Oosting J. Blood pressure response to dental checkup: a continuous, noninvasive registration. Gen Dent. 1991 Sep-Oct;39(5):339-42. No abstract available. PMID 1812051
- [Result] Gray RJ, Lomax AM, Rood JP. Periodontal ligament injection: with or without a vasoconstrictor? Br Dent J. 1987 Apr 11;162(7):263-5. doi: 10.1038/sj.bdj.4806100. No abstract available. PMID 3472559
- [Result] Grinberg M, Ávila WS, Amaral FMC. Modificações hemodinâmicas da gravidez. In: Andrade J, Ávila WS, editors. Doença cardiovascular, gravidez e planejamento familiar. São Paulo: Atheneu; 2003. p. 11-20.
- [Result] Haas DA, Pynn BR, Sands TD. Drug use for the pregnant or lactating patient. Gen Dent. 2000 Jan-Feb;48(1):54-60. PMID 11199555
- [Result] Hochman M, Chiarello D, Hochman CB, Lopatkin R, Pergola S. Computerized local anesthetic delivery vs. traditional syringe technique. Subjective pain response. N Y State Dent J. 1997 Aug-Sep;63(7):24-9. PMID 9297957
- [Result] Jastak JT, Yagiela JA. Vasoconstrictors and local anesthesia: a review and rationale for use. J Am Dent Assoc. 1983 Oct;107(4):623-30. doi: 10.14219/jada.archive.1983.0307. No abstract available. PMID 6355236
- [Result] Kim S. Ligamental injection: a physiological explanation of its efficacy. J Endod. 1986 Oct;12(10):486-91. doi: 10.1016/s0099-2399(86)80204-7. No abstract available. PMID 3465854
- [Result] Krochak M, Friedman N. Using a precision-metered injection system to minimize dental injection anxiety. Compend Contin Educ Dent. 1998 Feb;19(2):137-40, 142-3, 146 passim; quiz 150. PMID 9656861
- [Result] Kubo SH, Schulman S, Starling RC, Jessup M, Wentworth D, Burkhoff D. Development and validation of a patient questionnaire to determine New York Heart Association classification. J Card Fail. 2004 Jun;10(3):228-35. doi: 10.1016/j.cardfail.2003.10.005. PMID 15190533
- [Result] Lopes AC. Alterações anátomo-fisiológicas do sistema cardiocirculatório na gravidez. In: Lopes AC, Delascio D, editors. Cardiopatia e gravidez. São Paulo: Sarvier; 1986. p. 5-13.
- [Result] LUND A. Elimination of adrenaline and noradrenaline from the organism. Acta Pharmacol Toxicol (Copenh). 1951;7(4):297-308. doi: 10.1111/j.1600-0773.1951.tb02871.x. No abstract available. PMID 14894244
- [Result] Lund CJ, Donovan JC. Blood volume during pregnancy. Significance of plasma and red cell volumes. Am J Obstet Gynecol. 1967 Jun 1;98(3):394-403. No abstract available. PMID 5621454
- [Result] Malamed SF. Farmacologia dos anestésicos locais. In: Malamed SF, editor. Manual de anestesia local. Rio de Janeiro: Guanabara Koogan; 2001. p. 43-65.
- [Result] Malamed SF. Farmacologia dos vasoconstritores. In: Malamed SF, editor. Manual de anestesia local. Rio de Janeiro: Guanabara Koogan; 2001. p. 43-65.
- [Result] Malamed SF. Técnicas de injeção suplementares. In: Malamed SF, editor. Manual de anestesia local. Rio de Janeiro: Guanabara Koogan; 2001. p. 43-65.
- [Result] Malamed SF. The periodontal ligament (PDL) injection: an alternative to inferior alveolar nerve block. Oral Surg Oral Med Oral Pathol. 1982 Feb;53(2):117-21. doi: 10.1016/0030-4220(82)90273-0. PMID 6949113
- [Result] Mancia G, Bertinieri G, Grassi G, Parati G, Pomidossi G, Ferrari A, Gregorini L, Zanchetti A. Effects of blood-pressure measurement by the doctor on patient's blood pressure and heart rate. Lancet. 1983 Sep 24;2(8352):695-8. doi: 10.1016/s0140-6736(83)92244-4. PMID 6136837
- [Result] Mauri L, O'Gara PT. Valvular Heart Disease in the Pregnant Patient. Curr Treat Options Cardiovasc Med. 2001 Feb;3(1):7-14. doi: 10.1007/s11936-001-0080-z. PMID 11139785
- [Result] Meechan JG. Intraligamentary anaesthesia. J Dent. 1992 Dec;20(6):325-32. doi: 10.1016/0300-5712(92)90018-8. PMID 1452871
- [Result] Meyer FU. Haemodynamic changes under emotional stress following a minor surgical procedure under local anaesthesia. Int J Oral Maxillofac Surg. 1987 Dec;16(6):688-94. doi: 10.1016/s0901-5027(87)80054-1. PMID 3125267
- [Result] Meyer FU. Hemodynamic changes of local dental anesthesia in normotensive and hypertensive subjects. Int J Clin Pharmacol Ther Toxicol. 1986 Sep;24(9):477-81. PMID 3781681
- [Result] Moore PA. Selecting drugs for the pregnant dental patient. J Am Dent Assoc. 1998 Sep;129(9):1281-6. doi: 10.14219/jada.archive.1998.0425. PMID 9766109
- [Result] Morishima HO, Heymann MA, Rudolph AM, Barrett CT, James LS. Transfer of lidocaine across the sheep placenta to the fetus. Hemodynamic and acid-base responses of the fetal lamb. Am J Obstet Gynecol. 1975 Jul 1;122(5):581-8. doi: 10.1016/0002-9378(75)90053-8. PMID 1170757
- [Result] Mount GJ. A new classification and techniques for simple restorative dentistry. Ann R Australas Coll Dent Surg. 1998 Oct;14:94-8. PMID 10895619
- [Result] Mount GJ, Hume WR. A new cavity classification. Aust Dent J. 1998 Jun;43(3):153-9. doi: 10.1111/j.1834-7819.1998.tb00156.x. PMID 9707777
- [Result] Mount GJ, Hume WR. A revised classification of carious lesions by site and size. Quintessence Int. 1997 May;28(5):301-3. PMID 9452692
- [Result] Naftalin LW, Yagiela JA. Vasoconstrictors: indications and precautions. Dent Clin North Am. 2002 Oct;46(4):733-46, ix. doi: 10.1016/s0011-8532(02)00021-6. PMID 12436828
- [Result] Nahum GG, Uhl K, Kennedy DL. Antibiotic use in pregnancy and lactation: what is and is not known about teratogenic and toxic risks. Obstet Gynecol. 2006 May;107(5):1120-38. doi: 10.1097/01.AOG.0000216197.26783.b5. PMID 16648419
- [Result] Naidoo DP, Desai DK, Moodley J. Maternal deaths due to pre-existing cardiac disease. Cardiovasc J S Afr. 2002 Jan-Feb;13(1):17-20. PMID 11875603
- [Result] Nakamura Y, Matsumura K, Miura K, Kurokawa H, Abe I, Takata Y. Cardiovascular and sympathetic responses to dental surgery with local anesthesia. Hypertens Res. 2001 May;24(3):209-14. doi: 10.1291/hypres.24.209. PMID 11409642
- [Result] Nusstein J, Claffey E, Reader A, Beck M, Weaver J. Anesthetic effectiveness of the supplemental intraligamentary injection, administered with a computer-controlled local anesthetic delivery system, in patients with irreversible pulpitis. J Endod. 2005 May;31(5):354-8. doi: 10.1097/01.don.0000140565.88940.60. PMID 15851928
- [Result] Palatini P, Frigo G, Bertolo O, Roman E, Da Corta R, Winnicki M. Validation of the A&D TM-2430 device for ambulatory blood pressure monitoring and evaluation of performance according to subjects' characteristics. Blood Press Monit. 1998 Aug;3(4):255-260. PMID 10212363
- [Result] Partyka W, Pajszczyk-Kieszkiewicz T, Januszewicz-Witorzenc J, Swatko-Piotrowska K. [Effect of oral surgery on the fetus and uterus in complicated pregnancy]. Pol Tyg Lek. 1977 Aug 8;32(32):1245-7. No abstract available. Polish. PMID 896583
- [Result] Robson SC, Hunter S, Boys RJ, Dunlop W. Serial study of factors influencing changes in cardiac output during human pregnancy. Am J Physiol. 1989 Apr;256(4 Pt 2):H1060-5. doi: 10.1152/ajpheart.1989.256.4.H1060. PMID 2705548
- [Result] Rosner B. Fundamentals of biostatistics. 2nd ed. Boston: PWS Publishers; 1986. p. 584.
- [Result] SHIP II. The response of systolic and diastolic blood pressures to dental stress. Oral Surg Oral Med Oral Pathol. 1960 Apr;13:499-507. doi: 10.1016/0030-4220(60)90355-8. No abstract available. PMID 14446037
- [Result] Silberman SL, Cohen LA, Meydrech EF. Dental anxiety and needs in low-income pregnant women. Community Dent Oral Epidemiol. 1980 Apr;8(2):114-5. doi: 10.1111/j.1600-0528.1980.tb01268.x. PMID 6934058
- [Result] Siu SC, Sermer M, Harrison DA, Grigoriadis E, Liu G, Sorensen S, Smallhorn JF, Farine D, Amankwah KS, Spears JC, Colman JM. Risk and predictors for pregnancy-related complications in women with heart disease. Circulation. 1997 Nov 4;96(9):2789-94. doi: 10.1161/01.cir.96.9.2789. PMID 9386139
- [Result] Silversides CK, Colman JM, Sermer M, Siu SC. Cardiac risk in pregnant women with rheumatic mitral stenosis. Am J Cardiol. 2003 Jun 1;91(11):1382-5. doi: 10.1016/s0002-9149(03)00339-4. No abstract available. PMID 12767443
- [Result] Smith JH, Dawes GS, Redman CW. Low human fetal heart rate variation in normal pregnancy. Br J Obstet Gynaecol. 1987 Jul;94(7):656-64. doi: 10.1111/j.1471-0528.1987.tb03170.x. PMID 3620414
- [Result] Szekely P, Turner R, Snaith L. Pregnancy and the changing pattern of rheumatic heart disease. Br Heart J. 1973 Dec;35(12):1293-303. doi: 10.1136/hrt.35.12.1293. No abstract available. PMID 4759927
- [Result] Thornburg KL, Jacobson SL, Giraud GD, Morton MJ. Hemodynamic changes in pregnancy. Semin Perinatol. 2000 Feb;24(1):11-4. doi: 10.1016/s0146-0005(00)80047-6. PMID 10709851
- [Result] Timm NH. Multivariate analysis with applications in education and psychology. Monterrey: CA Brooks/Cole; 1975.
- [Result] Trierweiler MW, Freeman RK, James J. Baseline fetal heart rate characteristics as an indicator of fetal status during the antepartum period. Am J Obstet Gynecol. 1976 Jul 1;125(5):618-23. doi: 10.1016/0002-9378(76)90783-3. PMID 937386
- [Result] Ueland K, Metcalfe J. Circulatory changes in pregnancy. Clin Obstet Gynecol. 1975 Sep;18(3):41-50. doi: 10.1097/00003081-197509000-00007. No abstract available. PMID 1157366
- [Result] van Mook WN, Peeters L. Severe cardiac disease in pregnancy, part I: hemodynamic changes and complaints during pregnancy, and general management of cardiac disease in pregnancy. Curr Opin Crit Care. 2005 Oct;11(5):430-4. doi: 10.1097/01.ccx.0000179807.15328.f0. PMID 16175029
- [Result] van Mook WN, Peeters L. Severe cardiac disease in pregnancy, part II: impact of congenital and acquired cardiac diseases during pregnancy. Curr Opin Crit Care. 2005 Oct;11(5):435-48. doi: 10.1097/01.ccx.0000179806.15328.b9. PMID 16175030
- [Result] Villablanca AC. Heart disease during pregnancy. Which cardiovascular changes are normal or transient? Postgrad Med. 1998 Oct;104(4):183-4, 187-92. doi: 10.3810/pgm.1998.10.460. PMID 9793564
- [Result] Villablanca AC. Heart disease during pregnancy. Which cardiovascular changes reflect disease? Postgrad Med. 1998 Nov;104(5):149-56. doi: 10.3810/pgm.1998.11.407. PMID 9823391
- [Result] Vonesh EF, Schork MA. Sample sizes in the multivariate analysis of repeated measurements. Biometrics. 1986 Sep;42(3):601-10. PMID 3567293
- [Result] Walton RE, Abbott BJ. Periodontal ligament injection: a clinical evaluation. J Am Dent Assoc. 1981 Oct;103(4):571-5. doi: 10.14219/jada.archive.1981.0307. PMID 6945341
- [Result] Wood M, Reader A, Nusstein J, Beck M, Padgett D, Weaver J. Comparison of intraosseous and infiltration injections for venous lidocaine blood concentrations and heart rate changes after injection of 2% lidocaine with 1:100,000 epinephrine. J Endod. 2005 Jun;31(6):435-8. doi: 10.1097/01.don.0000148146.10314.1a. PMID 15917682
- [Result] Yagiela JA. Intravascular lidocaine toxicity: influence of epinephrine and route of administration. Anesth Prog. 1985 Mar-Apr;32(2):57-61. PMID 3859230
- [Result] Yagiela JA, Duffin SR, Hunt LM. Drug interactions and vasoconstrictors used in local anesthetic solutions. Oral Surg Oral Med Oral Pathol. 1985 Jun;59(6):565-71. doi: 10.1016/0030-4220(85)90181-1. PMID 3892411
- See also: One is about a InterNet Portal where it is possible to have access teses in the complete one, defended in all the University of Sao Paulo. — http://www.teses.usp.br/teses/disponiveis/5/5131/tde-18042007-090959